CLINICAL TRIAL: NCT04982042
Title: Outpatient and Home Pulmonary Rehabilitation Program for Post COVID-19 Patients
Brief Title: Post COVID-19 Pulmonary Rehabilitation Program
Acronym: COVID19REHAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário de Anapolis (Other)
Responsible Party: Principal Investigator, Luis Vicente Franco de Oliveira, Principal investigator, Centro Universitário de Anapolis
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID-19 PULMONARY REHAB
Record Dates: First submitted 2021-07-08; First posted 2021-07-29 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Covid19; COVID-19 Respiratory Infection; Lung Diseases; Respiratory Insufficiency; Muscle Weakness; Anxiety Disorder; Mixed With Depression (Mild)
Keywords: COVID-19; Pulmonary Rehabilitation; Pulmonary Function; Respiratory Physiotherapy; Respiratory Insufficiency
MeSH Terms: conditions — COVID-19; Lung Diseases; Respiratory Insufficiency; Muscle Weakness; Anxiety Disorders; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: To compare the effects of an Outpatient and Home Pulmonary Rehabilitation Program aimed at patients with pulmonary sequelae resulting from COVID-19 and with other chronic lung diseases on clinical symptoms, level of physical activity, functional status, quality of life, survival and in health maintenance costs by the government.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blinded to the data due to the fact that we have a group of patients undergoing the Outpatient Rehabilitation Program and another group of patients undergoing the Home Rehabilitation Program with follow-up by Tele-Rehabilitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post COVID-19 Outpatient Pulmonary Rehabilitation Program (Experimental): The outpatient Pulmonary Rehabilitation Program will be carried out at the Pulmonary Rehabilitation Laboratory, consisting of a combination of aerobic and strengthening exercises, lasting 12 weeks, with a frequency of 3 times a week, always in the morning. Each session consists of active warm-up exercises, upper and lower limb strengthening, aerobic conditioning and stretching exercises. The warm-up phase consists of intercalated calisthenic exercises for different muscle groups, according to each patient's tolerance.
  Interventions: Other: Pulmonary Rehabilitation
- Post COVID-19 Home Pulmonary Rehabilitation Program (Active Comparator): The Home Pulmonary Rehabilitation Program will be carried out at the patients' homes, consisting of the same combination of aerobic and strengthening exercises, lasting 12 weeks, 3 times a week, always in the morning. Each session consists of active warm-up exercises, upper and lower limb strengthening, aerobic conditioning and stretching exercises. The warm-up phase consists of intercalated calisthenic exercises for different muscle groups, according to each patient's tolerance. Patients will be monitored weekly via whatsapp.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — The Pulmonary Rehabilitation Program consists of a combination of aerobic and strengthening exercises, lasting 12 weeks, with a frequency of 3 times a week, always in the morning. Each session consists of active warm-up exercises, upper and lower limb strengthening, aerobic conditioning and stretching exercises. The warm-up phase consists of intercalated calisthenic exercises for different muscle groups, according to each patient's tolerance.

SUMMARY:
Coronavirus-2019 disease (COVID-19) is a highly infectious respiratory disease that causes respiratory, physical and psychological dysfunction in patients.

With the increased understanding of the severity of COVID-19 and clinical evidence in accordance with the opinions of first-line clinical experts involved in the treatment of this epidemic, the investigators believe that the participation of patients with sequelae of COVID-19 in a Pulmonary Rehabilitation Program would be of utmost importance.

According to recent scientific recommendations for patients with sequelae of COVID-19, respiratory rehabilitation would alleviate symptoms of dyspnea, anxiety and depression and, eventually, improve physical functions and quality of life.

Therefore, it is essential to anticipate early rehabilitation after the acute phase of ARDS, in order to limit the severity of the effects of the ICU and promote rapid functional recovery. Physiotherapy will play a role in providing exercise, mobilization and rehabilitation interventions for survivors of critical illnesses associated with COVID-19, in order to enable a functional social return.

DETAILED DESCRIPTION:
The investigatores propose a clinical, prospective and consecutive study composed of participants with pulmonary sequelae of COVID-19 and pulmonary diseases such as COPD, Asthma, Bronchitis, Emphysema, Bronchiectasis and pulmonary fibrosis. Initially, all patients will undergo a physical assessment, pulmonary function tests and nutritional assessment, in addition to applying the modified dyspnea scale of the MMRC (Modified Medical Research Council) and the 6-minute walk test (6MWT), according to the standards recommended by the American Thoracic Society (ATS).

The proposed Outpatient and Home Pulmonary Rehabilitation Program is based on the Guidelines recommended by the Brazilian Society of Pulmonology (SBPT) and by the Global Initiative for Chronic Obstructive Lung Disease (GOLD), with a minimum duration of 12 weeks, frequency of 3 weekly sessions, accompanied by health professionals in this field.

Patients who seek care at municipal and state health services in the city of Anápolis, (Goiás) will be recruited. Patients with clinically stabilized COVID - 19 sequelae will be considered eligible, and who agree to participate in the study, signing the Informed Consent .

The outpatient PRP consisted of a combination of aerobic and strengthening exercises, lasting 12 weeks, frequency 3 times a week. Each session will consist of active warm-up exercises, upper and lower limb strengthening, aerobic conditioning and stretching exercises. The warm-up phase consists of intercalated calisthenic exercises for different muscle groups, according to each patient's tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pulmonary sequelae post COVID-19
* Patients clinically stabilized
* Who agreed to participate in the clinical study, signing the informed consent form, will be considered eligible.

Exclusion Criteria:

* Hospitalized patients
* Patients who present clinical instability
* Patients who do not commit to adhering to the Pulmonary Rehabilitation Program

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Functional status after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on levels of functional status assessed with the Medical Research Council (MRC) Scale in patients with pulmonary sequelae resulting from COVID-19.
Exercise capacity after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on exercise capacity assessed with the six minutes Walk Test ( 6MWT) in patients with pulmonary sequelae resulting from COVID-19.

SECONDARY OUTCOMES:
Forced Vital Capacity after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on the forced vital capacity (FVC) measured by spirometry in patients with pulmonary sequelae resulting from COVID-19.
Forced Expiratory Volume in first second after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on the forced expiratory volume in first second (FEV1) measured by spirometry in patients with pulmonary sequelae resulting from COVID-19.
Inspiratory muscle strength after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on the inspiratory muscles strength measured by vacuometry in patients with pulmonary sequelae resulting from COVID-19.
Peripheral muscle strength after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on the peripheral muscle strength measured by Hand Grip Dynamometer in patients with pulmonary sequelae resulting from COVID-19.
Levels of anxiety and depression after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on the Anxiety and depression levels measured by the Hospital Anxiety and Depression scale in patients with pulmonary sequelae resulting from COVID-19.
Quality of Life after Pulmonary Rehabilitation Program (COVID-19REHAB) | 12 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on the Quality of Life levels measured by Medical Outcomes Study/SF-36 Questionnaire in patients with pulmonary sequelae resulting from COVID-19.
Health costs after COVID - 19. | 36 weeks
  Effects of an Ambulatory and Home Pulmonary Rehabilitation Program on healthcare costs verified through the financial expenses of patients with pulmonary sequelae resulting from COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Luis VF OLiveira, PhD, Principal Investigator — Evangelical University of Goiás - UNIEVANGELICA
Locations (1):
- Centro Universitário de Anápolis - UniEVANGÉLICA, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Clinical and demographic data of patients involved in this study will be made available to other researchers as requested.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After 02 years
Access Criteria: The clinical and demographic data of the patients involved in this study will be made available to other researchers as requested after the end of the study and for an indefinite period.
URL: https://www4.unievangelica.edu.br/ppg/movimento-humano-e-reabilitacao/laboratorios

REFERENCES:
- See also: This is the link to the Pulmonary Rehabilitation Laboratory where this clinical study will be developed. — https://www4.unievangelica.edu.br/ppg/movimento-humano-e-reabilitacao/laboratorios